CLINICAL TRIAL: NCT03229525
Title: Narrative Exposure Based Intervention For Post-Traumatic Stress Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Michael J. Telch, Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-06-0063
Record Dates: First submitted 2017-07-19; First posted 2017-07-25 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trauma Related Expressive Writing (Active Comparator): Participants randomized to this condition will complete six sessions during which they will write about their trauma for 20 minutes. The participant will receive instructions to write about the traumatic event that they feel affects them the most. For each session they will be instructed to write about the same event. For the first session, participants will complete psychoeducation and treatment rationale modules. The instructions for writing about the traumatic event will emphasize the importance of exploring their deepest emotions and thoughts at the time of the event, as well as providing detailed information about the event itself. For the remaining five writing sessions participants will be instructed to write about the same event and to focus on providing a detailed description of the part of the event that was most distressing to them, as well as how the event had affected their lives. A researcher will review the writing independently to ensure treatment compliance.
  Interventions: Behavioral: Trauma Related Expressive Writing
- Neutral Expressive Writing (Sham Comparator): Participants randomized to this condition will complete six sessions during which they will write about their day, without describing emotions or opinions. Previous research has shown a significant reduction of symptoms with this type of control writing condition in participants with PTSD (Sloan et al., 2011). A researcher will review the writing to ensure compliance.
  Interventions: Behavioral: Neutral Expressive Writing

INTERVENTIONS:
Behavioral: Trauma Related Expressive Writing — Participants will write about the traumatic event over the course of six sessions.
  Arms: Trauma Related Expressive Writing
Behavioral: Neutral Expressive Writing — Participants will write about a neutral event over the course of six sessions.
  Arms: Neutral Expressive Writing

SUMMARY:
Post-traumatic Stress Disorder (PTSD) is a debilitating mental disorder that affects approximately 7% of the general population. This project's aim is to develop a greater understanding of the efficacy and underlying mechanisms of narrative exposure based treatments for PTSD. Adult participants (N=162) who meet DSM-5 criteria for PTSD will be enrolled in a 3-arm randomized clinical trial consisting of trauma-related expressive writing, trauma-related expressive speaking, or a factual expressive writing control condition. Treatments will be manualized and conducted entirely through the Qualtrics survey platform. Treatment will consist of six sessions, three per week over two weeks, taking place via the internet. Assessments will be conducted pre-treatment, post-treatment, and at 1-month follow-up in the lab. Assessments will be comprised of symptom self-report measures as well as two tasks completed in an eye tracker: a reading task to evaluate mechanisms underlying trauma narrative processing and a sentence production task to evaluate attentional shifts when producing verbal information

Specific Aims and Hypotheses:

1. Develop and test the relative efficacy of two cost-effective internet-based expressive trauma therapies (written vs. spoken) relative to a non-trauma writing control for PTSD. We hypothesize that both trauma-focused expressive therapies will achieve more favorable outcomes at posttreatment and follow-up on measures of PTSD and depression symptoms, posttraumatic growth, and quality of life compared to the writing control.
2. Conduct exploratory analyses testing baseline PTSD severity, depression severity, trauma type, time since trauma, and emotional engagement in moderating the differential effects of the selected expressive therapies.
3. Test the moderation of (1) active language processing with eye tracking (i.e. how long certain words are fixated on). (2) selected linguistic elements (i.e., frequency of emotional words, frequency of the pronoun "I"), (3) perceived self-efficacy to cope with trauma memories; (4) perceived threat appraisals associated with intrusive trauma memories on treatment outcome at follow-up. We hypothesize that (1) fewer and shorter fixations on ideographic (i.e. personally relevant) trauma words when reading the trauma narrative in the eye tracker will be associated with reductions in PTSD symptoms at follow-up. (2) increased use of emotional words over the course of writing sessions will be associated with reductions in PTSD and depression symptoms at follow-up; (3) pre- to posttreatment increases in trauma memory acceptance self-efficacy; and (4) pre- to posttreatment reductions in trauma memory threat appraisals will be associated with greater symptom reduction at the follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between the ages of 18 and 65
2. Meets Diagnostic and Statistical Manual 5 criteria for PTSD
3. Able to give consent
4. Access to a computer in a private place
5. Completes initial writing samples online

Exclusion Criteria:

1. Impaired vision
2. Bipolar Disorder
3. Psychosis
4. Suicidality
5. Current trauma related treatment
6. Psychotropic medication <2 months or not stable (dosage variable) in past 2 months
7. Reading grade level > 6th grade level
8. Obsessive Compulsive Disorder
9. Traumatic Brain Injury

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change in PTSD symptom severity | Pre-treatment (baseline), Post-treatment (2-weeks), Follow-up (1 month, 3 months, 6 months)
  PTSD Symptom Checklist at each assessment
Change in Depression symptoms | Pre-treatment (baseline), Post-treatment (2-weeks), Follow-up (1 month)
  Becks Depression Inventory at each assessment
Change in Posttraumatic Growth | Pre-treatment (baseline), Post-treatment (2-weeks), Follow-up (1 month)
  Post Traumatic Growth Inventory at each assessment
Change in Reading Task indices | Pre-treatment (baseline), Post-treatment (2-weeks), Follow-up (1 month)
  Reading narratives in an eye tracker at each assessment
Change in Sentence Production Task indices | Pre-treatment (baseline), Post-treatment (2-weeks), Follow-up (1 month)
  Describing images in an eye tracker at each assessment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Telch, Phd, Principal Investigator — University of Texas at Austin; Mikael Rubin, MA, Study Director — University of Texas at Austin
Locations (1):
- Laboratory for the Study of Anxiety Disorders, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description Website for the Laboratory for the Study of Anxiety Disorders — http://utanxiety.com